CLINICAL TRIAL: NCT02003677
Title: A Trial Investigating the Pharmacokinetic and Pharmacodynamic Properties of FIAsp in Geriatric and Younger Adult Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3891; 2011-002626-46 (EudraCT Number); U1111-1121-8758 (Other: WHO)
Record Dates: First submitted 2013-11-28; First posted 2013-12-06 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp followed by NovoRapid® (Experimental): Each subject will be randomly allocated to a treatment sequence consisting of 2 dosing visits separated by a wash-out period of 3-12 days
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® followed by Insulin aspart (Active Comparator): Each subject will be randomly allocated to a treatment sequence consisting of 2 dosing visits separated by a wash-out period of 3-12 days
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Subjects - in a euglycaemic clamp setting - will receive a single dose. The trial products will be administered subcutaneously (s.c. under the skin).
  Arms: FIAsp followed by NovoRapid®
Drug: insulin aspart — Subjects - in a euglycaemic clamp setting - will receive a single dose. The trial products will be administered subcutaneously (s.c. under the skin).
  Arms: NovoRapid® followed by Insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetic (the exposure of the trial drug in the body) and pharmacodynamic (the effect of the investigated drug on the body)properties of FIAsp (faster-acting insulin aspart) in geriatric and younger adult subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-35 years (both inclusive) (younger adult group) or below or equal to 65 years (geriatric group) at the time of signing informed consent
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index (BMI) 18.5-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-11-29 (Actual); Primary Completion 2014-08-14 (Actual); Study Completion 2014-08-14 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 12 hours

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours
Maximum observed serum insulin aspart concentration | From 0 to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. Faster Onset and Greater Early Exposure and Glucose-Lowering Effect with Faster-Acting Insulin Aspart vs. Insulin Aspart: A Pooled Analysis in Subjects with Type 1 Diabetes. Diabetes. 2016; Suppl. 1: A239. doi:10.2337/db16-861-1374 http://dx.doi.org/10.2337/db16-861-1374
- [Result] Heise T, Hovelmann U, Zijlstra E, Stender-Petersen K, Jacobsen JB, Haahr H. A Comparison of Pharmacokinetic and Pharmacodynamic Properties Between Faster-Acting Insulin Aspart and Insulin Aspart in Elderly Subjects with Type 1 Diabetes Mellitus. Drugs Aging. 2017 Jan;34(1):29-38. doi: 10.1007/s40266-016-0418-6. PMID 27873152
- [Result] Haahr H, Pieber TR, Mathieu C, Gondolf T, Shiramoto M, Erichsen L, Heise T. Clinical Pharmacology of Fast-Acting Insulin Aspart Versus Insulin Aspart Measured as Free or Total Insulin Aspart and the Relation to Anti-Insulin Aspart Antibody Levels in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2019 May;58(5):639-649. doi: 10.1007/s40262-018-0718-6. PMID 30402720
- [Derived] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com